CLINICAL TRIAL: NCT06078215
Title: CERebrolysine Effect on Blood-brain Barrier / Endothelium Integrity During Reperfusion Therapy of acUte Ischemic Stroke (CERBERUS Study)
Brief Title: CERebrolysine Effect on Blood-brain Barrier in acUte Ischemic Stroke
Acronym: CERBERUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 392/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; blood-brain barrier; cerebrolysin
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin; Receptors, Tumor Necrosis Factor, Type I

STUDY DESIGN:
Intervention Model Description: A prospective longitudinal study will be performed in ischemic stroke patients who:
  1. are included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy - control (group A),
  2. are included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy plus Cerebrolysin (group B)
  3. are not referred to reperfusion therapy nor Cerebrolysin (group C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thrombolysis and/or mechanical thrombectomy (No Intervention): patients included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy - comparator
- Cerebrolysin (Experimental): patients included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy and treated with Cerebrolysin
  Interventions: Combination Product: Cerebrolysin
- No reperfusion therapy / no cerebrolysin (No Intervention): patients not referred to reperfusion therapy nor Cerebrolysin

INTERVENTIONS:
Combination Product: Cerebrolysin — Intravenous infusion of 30 ml Cerebrolysine in 500 ml of buffered crystalloid solution intravenously initiated within 12 hours from symptoms onset
  Other Names: FPF (Fine Particle Fraction)-1070
  Arms: Cerebrolysin

SUMMARY:
The study investigates whether Cerebrolysin stabilizes blood-brain barrier integrity in a manner that can be monitored using serum levels of the principal tight junction proteins, e.g., occludin (OCL), claudin-5 (CLN), and zonula occludens-1 (ZO-1), or other molecules known to be involved in BBB degradation, e.g., S100B and whether it protects against hemorrhagic transformation in ischemic stroke patients after reperfusion therapy (i.e. thrombolysis and/or mechanical thrombectomy).

DETAILED DESCRIPTION:
Hemorrhagic transformation (HT) of ischemic stroke can be identified in 3-40% of patients. The incidence varies depending on the definition used and the studied population. The severity of HT can be described using clinical and radiological tools and classified as asymptomatic/symptomatic, according to European Cooperative Acute Stroke Study classification and Heidelberg Bleeding Classification. Breakdown of the blood-brain barrier (BBB) is associated with an increased risk of developing a hemorrhagic transformation (HT) of ischemic stroke. In patients who received reperfusion therapy (thrombolysis, mechanical thrombectomy), secondary HT had a negative influence on the clinical course and outcome.

Tight junction (TJ) proteins are important cell adhesion components that stabilize endothelium cells lining and are responsible for maintaining the BBB integrity.

Biomarkers of BBB damage that can be evaluated during the early phases of stroke might be useful for predicting the risk of HT. Such biomarkers could also facilitate the decision of whether to begin thrombolytic therapy in acute ischemic stroke patients. Experimental data support the evidence for protective effect of Cerebrolysin on BBB integrity. Moreover, it diminished and reversed negative effect of recombinant tissue plasminogen activator (rtPA) used as thrombolytic agent on endothelial cells integrity. Cerebrolysin stabilized tight junction proteins expression: occludin, claudin-5 and zona occludens 1 (ZO1). In our previous study we have found that circulating TJs predict HT in ischemic stroke patients. Clinically evident HTs were associated with increased concentrations of occludin and S100B, an increase in the claudin-5/ZO-1 ratio, and a decreased level of vascular endothelial growth factor (VEGF). Claudin-5 levels also correlated with HT occurrence when estimated within 3 hours of stroke onset. The protective effects of Cerebrolysin were already clinically evidenced, however there are no available studies using biomarkers of BBB.

Aim of the study

We aim to investigate whether Cerebrolysin stabilizes BBB integrity in a manner that can be monitored using serum levels of the principal TJ proteins, e.g., occludin (OCL), claudin-5 (CLN), and zonula occludens-1 (ZO-1), or other molecules known to be involved in BBB degradation, e.g., S100B and whether it protects against HT in ischemic stroke patients after reperfusion therapy.

Study design

A prospective longitudinal study will be performed in ischemic stroke patients who:

1. are included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy - control (group A),
2. are included for reperfusion therapy (intravenous thrombolysis and/or mechanical thrombectomy plus Cerebrolysin (group B)
3. are not referred to reperfusion therapy nor Cerebrolysin (group C).

All patients with NIHSS score > 8 will receive 30 ml Cerebrolysin in 500 ml of buffered crystalloid solution intravenously initiated within 12 hours from symptoms onset.

Whole blood samples will be withdrawn at the admission, then within 1 to 3 days after stroke onset and at 7th day after stroke onset or when the endpoint will be reached by the patient. Occludin, claudin 5 and ZO-1 concentrations will be analyzed by means of home-made enzyme-linked immunosorbent assay.

Endpoint will include clinical worsening (increase in the NIHSS by > 4 points), radiologically evident hemorrhage or radiologically evident brain edema at control CT performed within 1 to 3 days after stroke onset.

Standard head CT will be performed in all patients at the admission, within 1 to 3 days after stroke onset, after worsening of clinical status and additionally when the differentiation between hemorrhage and contrast staining will be required in thrombectomy patients. Hemorrhagic transformation of ischemic stroke will be classified according to Table 1.

Clinimetric evaluation of all patients will include NIHSS every day for 7 days and at day 30. Modified Rankin scale (mRS) will be evaluated at visit 1,2,3,4 and 5; Barthel index at visit 4 and 5 and Montreal Cognitive Assessment Test at visit 5.

All patents will undergo current American Heart Association Guidelines for the Early Management of Patients with Acute Ischemic Stroke.

Expected results It is expected that Cerebrolysin can stabilize blood-brain barrier in ischemic stroke patients treated with reperfusion therapies via remodelling of tight junction proteins between endothelial cells. Such an effect measured by the levels of circulating tight junction proteins can translate into prevention of hemorrhagic transformation. To summarize, Cerebrolysine can guard blood-brain barrier integrity in ischemic stroke (Cerberus effect).

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke patients
* informed consent

Exclusion Criteria:

* no informed consent
* primary or metastatic brain tumor
* brain abscess
* encephalitis
* localized inflammation
* sepsis
* autoimmune diseases of central or peripheral nervous system
* Cerebrolysin hypersensitivity / allergy
* epilepsy
* severe kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
National Institute of Health Stroke Scale | every day for 7 days after stroke onset
  National Institute of Health Stroke Scale; score range: 1-42; 1-4 - Minor stroke; 5-15 - Moderate stroke; 16-20 - Moderate to severe stroke; 21-42 - Severe stroke
National Institute of Health Stroke Scale | at day 30 after stroke onset
  National Institute of Health Stroke Scale; score range: 1-42; 1-4 - Minor stroke; 5-15 - Moderate stroke; 16-20 - Moderate to severe stroke; 21-42 - Severe stroke
Detection of hemorrhagic transformation [range o:1] | within 1 to 3 days after stroke onset, after worsening of clinical status by more than 4 points in NIHSS
  hemorrhagic transformation on head computerized tomography
Concentration of plasma occludin [ng/mL] | at the admission, within 1 to 3 days after stroke onset
  Occludin is an enzyme (EC 1.6) that oxidizes NADH (Nicotinamide adenine dinucleotide)
Concentration of plasma occludin [ng/mL] | at 7th day after stroke onset
  Occludin is an enzyme (EC 1.6) that oxidizes NADH (Nicotinamide adenine dinucleotide)
Concentration of plasma claudin 5 [ng/mL] | at the admission, within 1 to 3 days after stroke onset
  Claudins are small (20-24/27 kilodalton (kDa)) transmembrane proteins.
Concentration of plasma claudin 5 [ng/mL] | at 7th day after stroke onset
  Claudins are small (20-24/27 kilodalton (kDa)) transmembrane proteins.
Concentration of plasma ZO1 [ng/mL] | at the admission, within 1 to 3 days after stroke onset
  Zonula occludens-1 ZO-1, also known as Tight junction protein-1
Concentration of plasma ZO1 [ng/mL] | at 7th day after stroke onset
  Zonula occludens-1 ZO-1, also known as Tight junction protein-1

SECONDARY OUTCOMES:
Modified Rankin scale [range 0:6] | at the admission, within 1 to 3 days after stroke onset
  Modified Rankin scale; 0-2 - good functional outcome; 3-6 - poor functional outcome
Modified Rankin scale [range 0:6] | at 7th day after stroke onset
  Modified Rankin scale; 0-2 - good functional outcome; 3-6 - poor functional outcome
Modified Rankin scale [range 0:6] | at the 30th +/- 5 day after stroke onset
  Modified Rankin scale; 0-2 - good functional outcome; 3-6 - poor functional outcome
Modified Rankin scale [range 0:6] | at 90th +/- 5 day after stroke onset
  Modified Rankin scale; 0-2 - good functional outcome; 3-6 - poor functional outcome
Barthel Index for Activities of Daily Living (ADL) [range 0:100] | 30th +/- 5 day after stroke onset
  measures the degree of assistance required by an individual; 0-20 - total dependency, 21-60 - severe dependency, 61-90 - moderate dependency, 91-100 - slight dependency
Barthel Index for Activities of Daily Living (ADL) [range 0:100] | at the 90th +/- 5 day after stroke onset
  measures the degree of assistance required by an individual; 0-20 - total dependency, 21-60 - severe dependency, 61-90 - moderate dependency, 91-100 - slight dependency
Death [range 0:1] | within 90 days after stroke onset
  survival measure
Montreal Cognitive Assessment Test [range 0:30] | at the 90th +/-5 day after stroke onset
  the assessment of cognitive functions; 26-30 - normal cognition, 18-25 - mild cognitive impairment, 10-17 - moderate cognitive impairment, <10 - severe cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Michalak, Prof., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- University Hospital, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazmierski R, Michalak S, Wencel-Warot A, Nowinski WL. Serum tight-junction proteins predict hemorrhagic transformation in ischemic stroke patients. Neurology. 2012 Oct 16;79(16):1677-85. doi: 10.1212/WNL.0b013e31826e9a83. Epub 2012 Sep 19. PMID 22993287
- [Background] Poljakovic Z, Supe S, Ljevak J, Starcevic K, Peric I, Blazevic N, Krbot-Skoric M, Jovanovic I, Ozretic D. Efficacy and safety of Cerebrolysin after futile recanalisation therapy in patients with severe stroke. Clin Neurol Neurosurg. 2021 Aug;207:106767. doi: 10.1016/j.clineuro.2021.106767. Epub 2021 Jun 18. PMID 34214867
- [Background] Teng H, Li C, Zhang Y, Lu M, Chopp M, Zhang ZG, Melcher-Mourgas M, Fleckenstein B. Therapeutic effect of Cerebrolysin on reducing impaired cerebral endothelial cell permeability. Neuroreport. 2021 Mar 24;32(5):359-366. doi: 10.1097/WNR.0000000000001598. PMID 33661804
- [Background] Kassner A, Roberts T, Taylor K, Silver F, Mikulis D. Prediction of hemorrhage in acute ischemic stroke using permeability MR imaging. AJNR Am J Neuroradiol. 2005 Oct;26(9):2213-7. PMID 16219824
- [Background] Zhang Y, Chopp M, Zhang ZG, Zhang Y, Zhang L, Lu M, Zhang T, Winter S, Doppler E, Brandstaetter H, Mahmood A, Xiong Y. Cerebrolysin Reduces Astrogliosis and Axonal Injury and Enhances Neurogenesis in Rats After Closed Head Injury. Neurorehabil Neural Repair. 2019 Jan;33(1):15-26. doi: 10.1177/1545968318809916. Epub 2018 Nov 30. PMID 30499355
- [Background] Lang W, Stadler CH, Poljakovic Z, Fleet D; Lyse Study Group. A prospective, randomized, placebo-controlled, double-blind trial about safety and efficacy of combined treatment with alteplase (rt-PA) and Cerebrolysin in acute ischaemic hemispheric stroke. Int J Stroke. 2013 Feb;8(2):95-104. doi: 10.1111/j.1747-4949.2012.00901.x. Epub 2012 Sep 26. PMID 23009193